CLINICAL TRIAL: NCT03198117
Title: Huaier Granule for Prevention of Recurrence and Metastasis of Stage II and III NSCLC After Postoperative Adjuvant Chemotherapy: A Multicenter Randomized, Double-blind, Placebo-controlled Clinical Trial, Along With a Registration Study
Brief Title: Huaier Granule for Prevention of Recurrence and Metastasis of Stage II and III Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Qidong Gaitianli Medicines Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HE-201701
Record Dates: First submitted 2017-05-31; First posted 2017-06-23 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Huaier Granule (Experimental): Huaier Granule
  Interventions: Drug: Huaier Granule
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo
- No-treatment Control (No Intervention): patients refused any treatment

INTERVENTIONS:
Drug: Huaier Granule — a Chinese traditional medicine
  Arms: Huaier Granule
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This study including two parts，one part is a randomized clinical trial design，another part is a registration study.

DETAILED DESCRIPTION:
This study include a multicenter, randomized, controlled, double-blind, placebo-controlled post-market clinical trial and a registration study.

The randomized clinical trial included subjects (n =798) will be randomly divided into experimental (n = 532) and control groups (n =266) according to a random number table. Patients in the experimental group will receive Huaier Granule (20g/time, 3 times/d). Patients in the control group will receive placebo (20g/time, 3 times/d). The registration study plan to recruitment at least 300 patients.

The primary outcome measures is disease-free survival，secondary outcome measures is 2-year overall survivals, ECOG-performance status, Karnofsky performance score and tumor markers (CEA、CYFRA21-1、SCC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete resection who are at TNM (primary tumor, regional nodes, metastasis) stage II-Ⅲa, postoperative pathology confirmed for non-small cell lung cancer;
* Has completed four cycle standard solution of adjuvant chemotherapy, or refused to accept the postoperative adjuvant chemotherapy;
* Patients between 18 and 70 years old, no gender restriction;
* Eastern Cooperative Oncology Group (ECOG) PS of two or less;
* Before the start of the study, patient fully understands the study and is willing to sign the informed consent form;

Exclusion Criteria:

* Receiving adjuvant chemotherapy patients started greater than 24 weeks from surgical resection;
* Refused adjuvant chemotherapy patients started greater than 8 weeks from surgical resection;
* Suspected malignant pleural effusion;
* There is no clear pathological diagnosis;
* Combined with other cancer;
* Patient have a positive surgical margin;
* Accept other treatment for lung cancer of postoperative；
* Combined with severe idiopathic disease of liver, kidney and hematopoietic system;
* Combined psychosis or AIDS;
* Allergy to the test drug;
* Pregnant or lactating women;
* Participation in any other clinical trial within three months;
* Conditions that are considered not suitable for this study investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 2-year
  disease-free survival

SECONDARY OUTCOMES:
overall survivals | 2-year
  overall survivals
Quality of Life | 2-year
  Quality of Life-EORTC QLQ-C30
KPS | 2-year
  Karnofsky
ECOG-PS | 2-year
  ECOG-PS
CEA | 2-year
  tumor markers
CYFRA21-1 | 2-year
  tumor markers
SCC | 2-year
  tumor markers

CONTACTS AND LOCATIONS:
Overall Officials: guoping sun, doctor, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- Du Ying Ying, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No